CLINICAL TRIAL: NCT00880828
Title: A Single-Center, Prospective, Randomized, Active Controlled, Single Blind, Parallel Design, Three Arms Trial Comparing Two Different Cervical Collar Combine With Acetaminophen and Acetaminophen Along for the Treatment in Patient With Cervical Radiculopathy and Radicular Pain
Brief Title: Comparing Two Different Cervical Collars for the Treatment in Patient With Cervical Radiculopathy and Radicular Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Kuo-Sheng Hung, MD, PhD, Taipei medical University-Wan Fang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008WFCRC-02
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Cervical Radiculopathy; Radicular Pain; Acute Neck Pain; Cervicobrachial Pain
Keywords: Cervical Radiculopathy; Radicular Pain; Acute neck pain; Cervicobrachial pain; Far-infrared ray; FIR; Cervical collar; Cervical device; FIR Device
MeSH Terms: conditions — Radiculopathy | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): FIR cervical collar plus Acetaminophen
  Interventions: Other: FIR cervical collar with Acetaminophen
- B (Active Comparator): Conservative cervical collar plus Acetaminophen
  Interventions: Other: Conservative cervical collar with Acetaminophen
- C (Placebo Comparator): Acetaminophen only
  Interventions: Drug: Acetaminophen only

INTERVENTIONS:
Other: FIR cervical collar with Acetaminophen — FIR cervical collar with Acetaminophen QID/PRN for 4 weeks
  Arms: A
Other: Conservative cervical collar with Acetaminophen — Conservative cervical collar with Acetaminophen QID/PRN for 4 weeks
  Arms: B
Drug: Acetaminophen only — Acetaminophen QID/PRN for 4 weeks
  Arms: C

SUMMARY:
The primary objective of the study is to investigate the efficacy of device with far-infrared (FIR) irradiation in these patients with acute cervical radiculopathy.

DETAILED DESCRIPTION:
Acute neck pain is a relatively common experience that usually declines and disappears within a couple weeks. Some patients do not recover and with time develop chronic cervical pain and nerve root compression which may result in cervical radiculopathy.

Far-infrared (FIR) ray is one of the topics in energy medicine which is tremendously studied for the past few years. A variety of FIR applications showed an enhancement of beneficial effects on healing therapy, even though there is limited technical approach and systemic study placed on the theoretical study of FIR ceramics processing and the emissivity optimizing.

The evident difficulties in finding the appropriate cervical radiculopathy therapy initiated the current study. The aim of the study is to evaluate the efficacy of the FIR cervical collar in patients with long-lasting cervicobrachial pain; in whom the pain had a distribution that corresponded to a specific nerve root compression revealed by MRI or electrophysiological study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 20 years
* Cervical radiculopathy defined by neck pain irradiating to one arm with at least one of the following:

  1. Provocation by neck movements or sensory changes in one or more adjacent dermatomes or diminished deep tendon reflexes in the affected arm.
  2. Muscle weakness in one or more adjacent myotomes.
* Neck Disability Index (NDI) score greater than or equal to 10 points
* Visual analog scale (VAS) score for neck pain greater than or equal to 40mm
* C-spine X-ray signs judge by investigator
* Prolong Neck pain for one week or longer
* Written consent from patient

Exclusion Criteria:

* Serious somatic or psychiatric disease(s)
* History of spinal tumors or spinal infection
* Ongoing physical therapy within 4 weeks
* Cervical instability judge by investigator
* History of contact dermatitis or known allergic reaction to collar material
* Known allergic reaction to acetaminophen
* Any other clinical condition which, in the opinion of the principal investigator, would not allow completion of this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-04 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Mean of change from baseline in Neck Disability Index after 2 weeks of treatment | 4 weeks

SECONDARY OUTCOMES:
Mean of change from baseline in Neck Disability Index after 4 weeks of treatment | 4 weeks
Mean of change from baseline in Visual analog scale for neck pain after 2 and 4 weeks of treatment | 4 weeks
Mean of change from baseline in nerve conduction velocity (NCV) tests after 4 weeks of treatment | 4 weeks
Mean of change from baseline in Nerve Excitability Test (NET) after 2 and 4 weeks of treatment | 4 weeks
Compare with Acetaminophen consuming of each arm after 4 weeks of treatment | 4 weeks
Device-related serious adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Sheng Hung, MD, PhD, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan